CLINICAL TRIAL: NCT04492709
Title: A Fixed Sequence, Open-Label Study to Assess the Effect of Multiple Doses of AZD5718 on the Pharmacokinetics of Oral Midazolam (a CYP450 3A Probe) in Healthy Subjects
Brief Title: A Study to Assess the Effect of Multiple Doses of AZD5718 on Pharmacokinetics of Oral Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D7550C00011
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Disease
Keywords: AZD5718, CYP3A4 substrate, Drug-drug Interaction, Fixed sequence, Midazolam, Open-label, Pharmacokinetics
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Midazolam; AZD5718

STUDY DESIGN:
Intervention Model Description: Fixed sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The subjects will receive oral midazolam solution of 2 mg as a single dose on 2 occasions, 6 days apart (Days 1 and 7). The first dose will be prior to dosing with oral AZD5718 tablet and the second dose after five administrations of AZD5718 under fasted conditions.
  Interventions: Drug: Midazolam; Drug: AZD5718

INTERVENTIONS:
Drug: Midazolam — The subjects will receive single doses of midazolam solution 2 mg/mL orally on Day 1 alone in Treatment Period 1 and on Day 7 co-administered with oral AZD5718 tablet in Treatment Period 3.
Drug: AZD5718 — The subjects will receive oral AZD5718 tablet once daily starting on Day 2 to Day 6 in Treatment Period 2 and on Day 7 co-administered with midazolam in Treatment Period 3.

SUMMARY:
In clinical practice, AZD5718 will be co-administered with CYP3A substrates. Therefore, it is important to determine the impact of AZD5718 on the pharmacokinetics (PK) of CYP3A4 substrates. The primary objective of this study is to evaluate the effect of AZD5718 on the PK of midazolam, a known sensitive CYP3A4 substrate.

DETAILED DESCRIPTION:
This is a Phase 1, fixed sequence, open-label study in healthy subjects, performed at a single study center. This study will consist of 3 treatment periods to assess the PK of midazolam when administered alone and in combination with multiple doses of AZD5718.

The study will comprise:

* A screening period of maximum 28 days;
* Three treatment periods during which subjects will be resident from the day before first dosing (Day -1) until at least 24 hours after last dosing (Day 7); discharged on the morning of Day 8, and;
* A final Follow-up Visit within 5 to 7 days after the last administration of investigational medicinal product (IMP).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.
* Male subject must adhere to the contraception methods details.
* Have a body mass index between 18.5 and 30 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* History or presence of acute pulmonary insufficiency, marked neuromuscular respiratory weakness, obsessional states, phobic states, sleep apnea syndrome, or unstable myasthenia gravis.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at screening and/or on admission to the Clinical Unit, as judged by the Investigator, including:

  1. Alanine aminotransferase > 1.5 x upper limit of normal (ULN);
  2. Aspartate aminotransferase > 1.5 x ULN;
  3. Bilirubin (total) > 1.5 x ULN; and
  4. Gamma glutamyl transpeptidase > 1.5 x ULN.
* Any clinically significant abnormal findings in vital signs (blood pressure and pulse; supine) at screening and/or admission to the Clinical Unit, as judged by the Investigator.
* Any clinically significant abnormalities on 12-lead electrocardiogram at screening, as judged by the Investigator.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus antibody.
* Known or suspected Gilbert syndrome.
* Known or suspected history of drug abuse in the last 2 years, as judged by the Investigator.
* Has received another new chemical or biological entity within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator. History of hypersensitivity to drugs with a similar chemical structure or class to AZD5718 or known hypersensitivity to benzodiazepines or to any formulation excipients.
* Current smokers or those who have smoked or used nicotine products within the 3 months prior to screening.
* Positive screen for drugs of abuse or cotinine at screening or on admission to the study unit, or positive screen for alcohol on screening or on admission to the study unit.
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed (other than hormone-replacement therapy for females) or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the Investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator. Excessive intake of alcohol defined as the regular consumption of more than 24 g of alcohol per day for men or 12 g of alcohol per day for women.
* Involvement of any AstraZeneca, Parexel, or study site employee or their close relatives.
* Subjects who have previously received AZD5718.
* Subjects with history of lactose intolerance.
* Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Subjects who cannot communicate reliably with the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma peak concentration (Cmax) of midazolam | Day 1-Day 2 and Day 7-Day 8: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours (h) post-dose
  Comparison of Cmax calculated when midazolam alone and calculated when midazolam was taken together with AZD5718
Area under plasma concentration-time curve from time zero to infinity (AUCinf) of midazolam | Day 1-Day 2 and Day 7-Day 8: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 h post-dose
  Comparison of AUCinf calculated when midazolam alone and calculated when midazolam was taken together with AZD5718
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) of midazolam | Day 1-Day 2 and Day 7-Day 8: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 h post-dose
  Comparison of AUClast calculated when midazolam alone and calculated when midazolam was taken together with AZD5718
Time to reach maximum observed plasma concentration (tmax) of midazolam | Day 1-Day 2 and Day 7-Day 8: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 h post-dose
  Comparison of tmax calculated when midazolam alone and calculated when midazolam was taken together with AZD5718
Half-life (t1/2) of midazolam | Day 1-Day 2 and Day 7-Day 8: pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 h post-dose
  Comparison of t1/2 calculated when midazolam alone and calculated when midazolam was taken together with AZD5718
Plasma concentrations of AZD5718 | Day 2-Day 7: at trough and Day 7: 4 h post-dose
  AZD5718 Plasma concentrations will be evaluated at trough and also at the expected time of tmax

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious AEs | AE: From Day 1 to post-treatment follow-up visit (Day 13); SAE: From screening to post-treatment follow-up visit (Day 13)
  The number and percentage of subjects with AEs and the number of events including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal 12-lead electrocardiogram (ECG) | At screening and post-treatment follow-up visit (Day 13)
  12-lead resting ECG safety assessments if there are any abnormal findings or if the Investigator considers it is required for any other safety reason including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal physical examination | At screening, Day -1, Day 1, Day 4, Day 7, Day 8, and post-treatment follow-up visit (Day 13)
  Any new or aggravated clinically relevant abnormal medical physical examination finding compared to the baseline assessment including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal blood pressure (BP) | For approximately 6 weeks (from screening to post-treatment follow-up)
  Observed values and change from baseline value in systolic and diastolic BP including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal pulse rate | For approximately 6 weeks (from screening to post-treatment follow-up)
  Observed values and change from baseline value in pulse rate including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal oxygen saturation levels | On Day 1 and Day 7: 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8 and 12 h post-dose
  Observed values and change from baseline value in oxygen saturation including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal hematology parameters | At screening, Day -1, Day 1 (pre-dose), Day 2 and Day 4 (pre-dose), Day 7 (pre-dose), Day 8, and post-treatment follow-up visit (Day 13)
  Observed values and change from baseline value in hematology including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal clinical chemistry parameters | At screening, Day -1, Day 1 (pre-dose), Day 2 and Day 4 (pre-dose), Day 7 (pre-dose), Day 8, and post-treatment follow-up visit (Day 13)
  Observed values and change from baseline value in clinical chemistry including for both AZD5718 alone and in combination with midazolam
Number of subjects with abnormal urine analysis parameters | At screening, Day -1, Day 1 (pre-dose), Day 2 and Day 4 (pre-dose), Day 7 (pre-dose), Day 8, and post-treatment follow-up visit (Day 13)
  Observed values and change from baseline value in urine analysis including for both AZD5718 alone and in combination with midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Pablo Forte Soto, MD, MSc, PhD, Principal Investigator — Parexel Early Phase Clinical Unit London
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home